CLINICAL TRIAL: NCT03993470
Title: The Effects of Short-foot Exercises in the Foot Posture
Brief Title: The Effects of Short-foot Exercises in Foot Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Aurora Castro Mendez, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0465
Record Dates: First submitted 2019-06-13; First posted 2019-06-20 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Pronation Deformity of the Foot
Keywords: pronation

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): The short foot exercise daily for 4 weeks
  Interventions: Behavioral: Short foot excercise for intrinsec muscles of the foot
- Control (Placebo Comparator): A placebo excercise daily for 4 weeks
  Interventions: Behavioral: Short foot excercise for intrinsec muscles of the foot

INTERVENTIONS:
Behavioral: Short foot excercise for intrinsec muscles of the foot — to examine the effects of the SFE compared to a placebo exercise in the foot posture index after a daily period of 4 weeks.

SUMMARY:
Therefore, the aim of this study is to examine the effects of the short foot exercises compared to placebo exercises in the foot posture index after a daily period of 4 weeks.

DETAILED DESCRIPTION:
The intrinsic foot muscles collaborate in maintain the media longitudinal arch and in the postural control of the body.1 The plantar intrinsic foot muscles play a crucial role providing the foot stability and flexibility. 2 There are few studies about the relationship between hyperpronation and the training of the intrinsic muscles.

A specific training program as a "short foot exercise" (SFE) may improve pathological conditions involving the foot and the lower extremity including plantar fasciitis, tendinopathies and foot hiperpronation.3 Several balance training techniques have been applied for improving postural stability, and the SFE have been widely accepted by physiotherapists to improve the longitudinal arch foot and the body segments.4 In this study, the foot posture will be evaluated with the foot posture index (FPI) and the navicular drop test (NDT). The foot posture index is a validated and useful method like a complementary tool for evaluating foot disorders. 5. The foot posture quantify the foot posture as normal, pronated or supinated. The foot posture index indicates a pronated foot position in a support relaxed position when IPP is equal to or superior to a +6 value. 5 The Navicular Drop Test quantifies, in millimeters, the descent of the navicular tuberosity. It was developed to evaluate the pronation of the foot and, consequently, the drop of the medial longitudinal arch, a excessively pronated foot (NDT≥10mm).6.

Therefore, the aim of this study is to examine the effects of the SFE compared to a placebo exercise in the foot posture index after a daily period of 4 weeks.

There is a lack of evidence of the effect of training intrinsic muscles in foot posture.

The hypothesis of the researches is that the SFE may contribute to improving the pronated foot posture. This treatment may allow normalizing the foot posture and the kinematic interaction of the lower extremity joints during walking.

ELIGIBILITY:
Inclusion Criteria:

Males and females between 18 and 65 years old.

-

Exclusion Criteria:

* The exclusion criteria: serious illness, current participation in another research study, pregnancy, previous foot surgery, current treatment of foot pathology.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Foot posture index | four weeks
  the foot posture will be evaluated with the foot posture index (FPI) .The foot posture index is a validated and useful method like a complementary tool for evaluating foot disorders. 5. The foot posture quantify the foot posture as normal, pronated or supinated. A podiatrist assessed the foot posture during the biomechanical assessment based on the six-item foot posture index (FPI≥+6). The FPI consists of six validated items measured in a standing relaxed position of the subject; The categories are: Supinated foot: -1 a -12. Neutral foot posture: 0 to +5 (neutral). Pronated foot posture: +6 to +12.

CONTACTS AND LOCATIONS:
Overall Officials: aurora c castro mendez, Principal Investigator — Departament of Podiatry. University of Seville
Locations (1):
- Aurora Castro Mendez, Seville, Spain